CLINICAL TRIAL: NCT03136913
Title: A Comparison Between Primary and Secondary Flap Coverage in Extraction Sites: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Yong Hur, Assistant Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11441
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Loss of Teeth Due to Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Closed Flap Technique (Active Comparator): Healing by primary intention: Extraction and ridge preservation, utilizing non-resorbable membrane (Cytoplast® TXT-200 ) and freeze dried bone allograft (MinerOss® Cortical and Cancellous Chips (FDBA)), with flaps in primary coverage.
  Interventions: Device: Cytoplast® TXT-200; Device: MinerOss® Cortical and Cancellous Chips (FDBA); Procedure: Closed Flap Technique
- Open Flap Technique (Active Comparator): Healing by secondary intention: Extraction and ridge preservation, utilizing non-resorbable membrane (Cytoplast® TXT-200) and freeze dried bone allograft (MinerOss® Cortical and Cancellous Chips (FDBA)), with flaps in position for healing by secondary intention.
  Interventions: Device: Cytoplast® TXT-200; Device: MinerOss® Cortical and Cancellous Chips (FDBA); Procedure: Open Flap Technique

INTERVENTIONS:
Device: Cytoplast® TXT-200 — Non-resorbable membrane
Device: MinerOss® Cortical and Cancellous Chips (FDBA) — Mixture of allograft mineralized cortical and cancellous chips
Procedure: Open Flap Technique — After extraction, the socket wound is left open to heal by secondary intention
  Arms: Open Flap Technique
Procedure: Closed Flap Technique — After extraction, the socket wound is closed by primary closure
  Arms: Closed Flap Technique

SUMMARY:
This study is being conducted to compare the outcomes of two separate surgical techniques used in tooth extraction and ridge preservation. Ridge preservation is done to potentially minimize the amount of bone loss that occurs between the tooth extraction and implant or bridge placement, as compared to leaving the extraction site empty. There are two techniques that are commonly used for these procedures, either to close the surgical site of the extracted tooth with sutures (closed flap technique) or to leave the extraction site open to heal naturally (open flap technique). In the open flap technique there will be sutures used to secure and hold down the material used to cover the wound, called a non-resorbable membrane. The flaps will remain in their natural position, the site will fill up naturally with new tissue from the bottom up and then close itself in from the sides. The investigators want to see which technique offers better healing and reduces bone loss.

DETAILED DESCRIPTION:
Study design will be a single center, randomized controlled trial, split mouth designed study, to compare the bone dimensional changes following extraction and ridge preservation in surgical techniques that leave the flap open and closed.

The primary aim of this study is to evaluate the bone dimensional changes following extraction and ridge preservation with primary coverage (closed flap technique) in comparison to secondary intention (open flap technique).

The investigators hypothesize that the closed flap technique will have more potential to maintain vertical bone height when compared with the open flap technique, due to less susceptibility from infection and inflammation.

Secondary aim is to evaluate patients' self-report of postoperative discomfort. The investigators hypothesize that open flap technique will have less post-operative pain/discomfort due to less flap dissection and elevation when compared to closed flaps.

Tertiary aim is to have a histomorphometric examination and to assess the formation of new bone.

The investigators hypothesize that better bone volume percentage will be observed in closed flap technique when compared to open flap technique.

The primary outcome is the mean difference in alveolar bone height change between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is treatment planned at Tufts University School of Dental Medicine (TUSDM) for extraction and future implant placement and meet all medical and dental requirements of the TUSDM periodontology clinic for periodontal surgery (e.g., subjects with no diseases or medication allergies contraindicating periodontal surgery).

  * Patient must have bilateral extraction (canine to molar) sites of teeth located on the same arch (e.g. upper right and upper left) treatment planned for future implant placement at TUSDM.
  * The number of teeth planned for extraction (either one or two adjacent) and ridge preservation should match the same number of teeth (either one or two adjacent) from the contra-lateral side on the same arch.
  * Presence of at least 3 intact bony walls and at least half of the fourth bony wall at each site as determined by bone sounding at Visit 1.

Exclusion Criteria:

* Have any known disease that interferes with periodontal surgery and would not allow the patient to be treatment planned for the procedures in the TUSDM periodontology clinic (e.g., severe anemia, low white blood cell count, bleeding or coagulation disorder, uncontrolled hypertension (150/90), recent myocardial infarction (within 6 months of enrollment), diabetes (HbA1C ≥7%), HIV/AIDS (self-reported), history of or currently undergoing head and neck radiation, history of or currently taking bisphosphonates).

  * Subject who has a disease or condition that may affect hard and soft tissue healing (e.g., previous or current head and neck radiation therapy, long term steroid use defined as more than two weeks in the past two years).
  * Subject who has diseases that affect bone metabolism (e.g., osteoporosis, osteopenia).
  * Pregnancy (self-reported)
  * Current Smokers
  * Extraction socket with > 50% bone loss on the buccal or lingual/palatal bone as determined by bone sounding at Visit 1.
  * Allergic to gentamycin, povidone-iodine, or surfactants as trace amounts may be contained in the MinerOss®

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02-17 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Hur, DMD, MSc, Principal Investigator — TUSDM
Locations (1):
- Tufts University School of Dental Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aladmawy MA, Natto ZS, Kreitzer M, Ogata Y, Hur Y. Histological and histomorphometric evaluation of alveolar ridge preservation using an allograft and nonresorbable membrane with and without primary closure: A pilot randomized controlled clinical trial. Medicine (Baltimore). 2022 Jul 1;101(26):e29769. doi: 10.1097/MD.0000000000029769. PMID 35777057
- [Derived] Aladmawy MA, Natto ZS, Steffensen B, Levi P, Cheung W, Finkelman M, Ogata Y, Hur Y. A Comparison between Primary and Secondary Flap Coverage in Ridge Preservation Procedures: A Pilot Randomized Controlled Clinical Trial. Biomed Res Int. 2019 Aug 20;2019:7679319. doi: 10.1155/2019/7679319. eCollection 2019. PMID 31531367

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two randomization schemes were created using the statistical package R Version 2.11.1. One randomization scheme was used if the subject has more than 1 set of qualifying sites (the inclusion criteria specify bilateral sites) and randomized which set would be included in the study. The other randomization scheme was used to randomize which side is in Group 1 and which side is in Group 2. The two sites (one set) chosen to be in the study each had a 50% chance of being in either group.
Groups:
- All Study Participants (OFT vs CFT): Open flap technique (OFT) with secondary wound closure (test group) and closed flap technique (CFT) with primary wound closure (control group).
  OFT with flaps in position for healing by secondary intention CFT with flaps in primary coverage
Period: Overall Study
Arm/Group | All Study Participants (OFT vs CFT)
Started | 13
Subjects Received Both Intervention | 10 (10 subjects with 10 OFT and 10 CFT sites received clinical measurement before implant surgery)
Completed | 8 (8 subjects with 8 OFT and 8 CFT sites received implant surgery)
Not Completed | 5

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants (OFT vs CFT): Open flap technique (OFT) with secondary wound closure (test group) Closed flap technique (CFT) with primary wound closure (control group).
Arm/Group | All Study Participants (OFT vs CFT)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  gender: Female | 2
  gender: Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Alveolar Bone Height Change
Description: Models/casts will be made in stone using the impressions. A stent will be made to measure the height and width of the alveolar ridge. Ridge height will be measured before tooth extraction, and 3-5 months after ridge preservation.
Time Frame: < 6 months post extraction and ridge preservation
Population: 20 sites were analyzed of 10 participants, 10 OFT sites and 10 CFT sites, 1 OFT and 1 CFT for each subject, were analyzed
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: site
Groups:
- OFT vs CFT: Open flap technique (OFT) with secondary wound closure (test group) and closed flap technique (CFT) with primary wound closure (control group).
Arm/Group | OFT vs CFT
Number analyzed (Participants) | 10
Number analyzed (site) | 20
mm
  OFT | 7.5 (1.8)
  CFT | 8.1 (1.9)

2. Secondary Outcome: Post-operative Pain/Discomfort
Description: Subjects will be asked to rate their pain/discomfort on a visual analog scale (VAS) questionnaire (scores on a scale of 0-10, 10 to be the worst)
Time Frame: Up to 16 days post extraction and ridge preservation
Population: 10 subject received CFT and OFT simultaneously. Post-operative pain/discomfort comparing the two techniques were analyzed
Measure: Mean (Standard Deviation); unit: VAS(scale 0-10), scores on a scale
Arm/Group | Open Flap Technique | Closed Flap Technique
Number analyzed (Participants) | 10 | 10
VAS(scale 0-10), scores on a scale
  24 hours | 1.1 (0.5) | 3 (0.8)
  2 weeks | 0.4 (0.5) | 0.8 (0.9)

3. Secondary Outcome: Percentage New Bone Formation
Description: Histomorphometric analysis of bone core biopsy to determine percent new bone formation
Time Frame: Up to 6 months post extraction and ridge preservation
Population: 16 sites were analyzed of 8 participants, 8 OFT sites and 8 CFT sites were analyzed
Measure: Mean (Standard Deviation); unit: percentage of new bone formation
Units Other Than Participants: site
Arm/Group | Open Flap Technique | Closed Flap Technique
Number analyzed (Participants) | 8 | 8
Number analyzed (site) | 8 | 8
percentage of new bone formation | 34 (15) | 39 (10)

ADVERSE EVENTS:
Time Frame: None to report during the study period, 1 year.
Description: Adverse events were recorded in source documents and on case report forms. All adverse events and non-serious situations were recorded, monitored, and reported to the IRB at the time of continuing review or at the study's termination.
Groups:
- Open Flap Technique (OFT): Open flap technique (OFT, test group) with secondary wound closure
- Closed Flap Technique (CFT): closed flap technique (CFT, control group) with primary wound closure
Arm/Group | Open Flap Technique (OFT) | Closed Flap Technique (CFT)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No